CLINICAL TRIAL: NCT06224296
Title: The Exploratory Study About the Effect of Using Double Filtration Plasmapheresis (DFPP) Removing Inflammatory Cytokines, Lipids and Toxic Metal Ions in Peripheral Blood in Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Cell Therapy Group Co.,Ltd (Industry)
Collaborators: Shanghai Mengchao Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BZXJ2401-A-01
Record Dates: First submitted 2024-01-16; First posted 2024-01-25 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Sub-healthy; Hyperlipidemia; Toxic Metal Ions Accumulation
Keywords: DFPP; Blood Purification
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Intervention Model Description: Subjects are self-controlled in each group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A: Inflammatory cytokine group (Experimental): Self-control
  Interventions: Device: DFPP
- Group B: Lipid group (Experimental): Self-control
  Interventions: Device: DFPP
- Group C: Toxic metal ions group (Experimental): Self-control
  Interventions: Device: DFPP

INTERVENTIONS:
Device: DFPP — One session of blood purification using DFPP to remove inflammatory cytokines in peripheral blood.
  Arms: Group A: Inflammatory cytokine group
Device: DFPP — One session of blood purification using DFPP to remove lipids in peripheral blood.
  Arms: Group B: Lipid group
Device: DFPP — One session of blood purification using DFPP to remove toxic metal ions.
  Arms: Group C: Toxic metal ions group

SUMMARY:
This study investigates whether using Double Filtration Plasmapheresis (DFPP) could improve the overall health of adults through removing inflammatory cytokines, lipids and toxic metal ions from peripheral blood. It's also postulated that DFPP could boost immune cells through removing certain inflammatory cytokines and blood lipids.

DETAILED DESCRIPTION:
In this study, 3 groups of subjects will be recruited based on the indications of using DFPP. Estimated 100 sub-healthy subjects will be enrolled in the Group A (inflammatory cytokine group), the inflammatory cytokine panel will be tested at baseline, immediately and 1, 3, 6 months after using DFPP. Similarly estimated 100 subjects with elevated blood lipid or cholesterol will be enrolled in Group B (lipids group), the lipid panel will be tested at the same timeline as Group A. Estimated 50 subjects who are likely to have toxic metal ions accumulated (eg. using make-up for long term, working exposure) will be enrolled in Group C (toxic metal ions group), the specific metal ions will be tested before and after using DFPP. Tests related to immune cells will also be conducted in Group A and B at baseline, immediately and 1, 3, 6 months after using DFPP.

ELIGIBILITY:
Inclusion Criteria:

* Male/females of 18 to 85 years of age. For Group B, subjects should have elevated blood lipid or cholesterol, which could be a. hyperlipidemia; b. higher than the normal range but not high enough to be diagnosed as hyperlipidemia. Able to provide written Informed Consent. Able to follow verbal and written study directions.

Exclusion Criteria:

* Have sever liver and kidney dysfunction. Have cardiopulmonary insufficiency. Have solid or blood tumor. Pregnancy or breastfeeding women.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Inflammatory cytokine panel | Baseline, day0, 1, 3, 6 month after DFPP
  IL-2,IL-4,IL-6,IL-10, TNF-a, IFN-r, hs CRP(subjected to change)
Blood lipid panel | Baseline, day0, 1, 3, 6 month after DFPP
  Total cholesterol, total triglycerides, low-density lipoprotein(LDL), high-density lipoprotein(HDL), lipoprotein(a)(subjected to change)
Toxic metal ions | Baseline, day0
  Lead, mercury etc based on the specific exposure

SECONDARY OUTCOMES:
Immune cells | Baseline, day0, 1, 3, 6 month after DFPP
  TBNK, ROS, PD1/lag3/KLRG1/CD57 etc (subjected to change)

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mengchao Cancer Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No